CLINICAL TRIAL: NCT04142255
Title: A Clinical Study to Explore the Efficacy of Fecal Mircobiota Transplantation (FMT) in the Treatment of Childhood ASD Patients With Gastrointestinal Symptoms
Brief Title: Explore Efficacy of FMT Treating Childhood ASD Patients
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The review board rejected our request of changing the protocol and advised us to terminate the trial.
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XH-19-008
Record Dates: First submitted 2019-09-08; First posted 2019-10-29 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-08

CONDITIONS: ASD Accompanied by Moderate to Severe Gastrointestinal Symptoms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT (Experimental): 20 subjects will be enrolled in this arm to receive FMT treatment.
  Interventions: Biological: FMT

INTERVENTIONS:
Biological: FMT — FMT administration starts on the first week of enrollment. Age-based dose of FMT is taken once a day for the first three days of the first week. Then once a week for 3 weeks.

SUMMARY:
To explore the efficacy of fecal microbiota transplantation (FMT) in improving the gastrointestinal symptoms and autism symptoms in patients diagnosed as autism spectrum disorder (ASD) comorbid with gastrointestinal symptoms.

DETAILED DESCRIPTION:
This trial is designed to reconstruct the intestinal micro-ecology of children with ASD by the interventional treatment of FMT. At the same time, combined with metagenomics and 16S rRNA sequencing techniques, the trial aims to study the efficacy of intestinal micro-ecology for the treatment of autism symptoms and the improvement of gastrointestinal problems and autism symptoms in autistic patients, and to explore potential new techniques for treating children with ASD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with ASD. Diagnostic criteria: diagnosed by pediatric psychiatrists in accordance with the criteria in the Fifth Edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-V), Autism Diagnostic Observation Schedule (ADOS) and Autism Diagnostic Interview-Revised (ADI-R);
2. Patients with moderate to severe gastrointestinal symptoms which are not life-threatening and do not require immediate surgery;
3. Patients aged 3-17 years, male or female;
4. Patients who are suitable for receiving oral FMT capsules, and able to swallow the capsules without chewing;
5. Patients who are able to complete the study as required by the trial protocol;
6. Patients without known immunodeficiency diseases;
7. Subjects and/or their guardians are able to fully understand the informed consent of the trial, and voluntarily sign the informed consent form.

Exclusion Criteria：

1. Patients diagnosed with severe malnutrition;
2. Patients depend on tube feeding (liquid food);
3. Patients with a serious gastrointestinal disease requiring immediate treatment (or life-threatening);
4. Patients with primary immunodeficiency disease during screening;
5. Patients with a single-gene disorder;
6. Patients with a history of severe allergies;
7. Patients with severe fever and/or serious infection within 7 days prior to enrollment;
8. Patients with renal insufficiency and liver dysfunction (or creatinine > 2 mg/dl, direct bilirubin > 2 mg/dl);
9. Subjects with congenital or acquired immunodeficiency or immunosuppression (e.g., neoplastic disease or organ transplant) who have received or are undergoing chemotherapy, or have been diagnosed with HIV;
10. Patients with inflammatory bowel disease, celiac disease, large intestine irritation or eosinophilia, esophagitis, eosinophilic gastroenteritis or similar diseases;
11. Subjects with severe sensory or motor disorders (e.g., blindness, deafness, seizures, cerebral palsy);
12. Patients who are participating in other clinical studies, or have received interventions in other interventional clinical studies within 4 weeks prior to enrollment.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale (GSRS) | Baseline to 12 weeks
  The Gastrointestinal Symptom Rating Scale (GSRS) is an interview-based rating scale consisting of 15 items for assessment of bowel function, which refers to the period of the previous week and requires a short time to fill and has easy-to-understand questions on gastrointestinal symptoms. Changes in the Gastrointestinal Symptom Rating Scale (GSRS) before and after treatment.
Childhood Autism Rating Scale (CARS) | Baseline to 12 weeks
  The CARS is a 15-item measure that clinicians complete based on observations from the child and subsequent interviews with the caregivers.The total score on the CARS reflects the symptom level of ASD with lower scores indicating minimal ASD symptoms and higher scores representing severe ASD symptoms. Changes in the Childhood Autism Rating Scale (CARS) before and after treatment.

SECONDARY OUTCOMES:
Daily Stool Records (DSR) | From the treatment period to Week 12
  The Daily Stool Records (DSR) is a self-designed questionaire to record each participant's stool per day during the study. Changes in the Daily Stool Records (DSR) before and after treatment.
Safety and Tolerability | Baseline to 12 weeks
  Safety and Tolerability refer to treatment-related adverse events as assessed by CTCAE v5.0 in the 12-week observation after the treatment.
Developmental Quotient/Intelligence Quotient Scale (DQ/IQ) | Baseline to 12 weeks
  The (DQ/IQ) is evaluated by specialists in an intelligence test designed for children. Three versions of the intelligence test are the Gesell Developmental Schedules, the Wechsler Preschool and Primary Scale of Intelligence (WPPSI) and the Wechsler Intelligence Scale for Children-Revised (WISC-R), which are selected according to each participant's age. Changes in the Developmental Quotient/Intelligence Quotient Scale (DQ/IQ) before and after treatment.
Autism Diagnostic Observation Schedule (ADOS) | Baseline to 12 weeks
  The ADOS is a structured play session conducted by clinicians, which includes a series of social communication and play "presses" to diagnose ASD. For younger children, social interest, joint attention, communication, symbolic play, and repetitive behaviors are assessed. Changes in the Autism Diagnostic Observation Schedule (ADOS) before and after treatment.
Social Responsiveness Scale (SRS) | Baseline to 12 weeks
  The SRS measures the severity of social interaction impairments in ASD populations, sensitive between 3 to 18 years of age.It provides an impression of observed social impairments, assessing domains of communication, social interactions, and repetitive and stereotyped behaviors and interests. Changes in the Social Responsiveness Scale (SRS) before and after treatment.
Clinical Global Impressions-Improvement (CGI-I) Scale | Baseline to 12 weeks
  The CGI-I assesses how much the patient's condition has improved or worsened relative to a baseline state, ranging from 1 (very much improved) to 7 (very much worse), and is recommended for all clinical trials involving participants with ASD.Improvement was defined as a score of 3 (minimally improved) or lower. Changes in the Clinical Global Impressions-Improvement (CGI-I) Scale before and after treatment.
Long Term Safety Assessed Through Adverse Events | [16, 20, 24 weeks]
  Long Term Safety refers to treatment-related as assessed by CTCAE v5.0 after the 12-week study. Evaluation of safety telephone follow-up after 12 weeks.

OTHER OUTCOMES:
Head Magnetic resonance imaging (MRI) | Baseline to 12 weeks
  Head MRI is used to detect the structure of the brain. Changes in the head MRI results of the subject before and after treatment.
Children's Dietary Diversity Questionnaire | Baseline to 12 weeks
  Children's Dietary Diversity Questionnaire is a scale consisting of 8 categories of food each scoring from 0 to 2 based on the frequency. Changes in the subject's dietary diversity questionnaire results before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, Professor, Principal Investigator — Xinhua hospital Affilated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- ShanghaiXinhua, Shanghai, Shanghai Municipality, China